CLINICAL TRIAL: NCT03195439
Title: Temple Touch Pro (TTP) Non-Invasive Core Temperature Monitoring as a Measure for Early Detection of Fever Related Infections, Including Sepsis.
Acronym: TTP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medisim Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0068-17
Record Dates: First submitted 2017-06-12; First posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Patients in ICU

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients in ICU (Experimental)
  Interventions: Device: TTP

INTERVENTIONS:
Device: TTP — TTP™ allows to continuously measure body temperature using a new non-invasive method, and was cleared for marketing by US FDA (K150160) for as a temperature monitoring system intended to measure and monitor core body temperature of patients of all ages, by applying a sensor unit on the forehead.

SUMMARY:
The study has 2 phases:

* The Retrospective Phase (50 patients were diagnosed to have sepsis according to our definition and criteria and 30 patients as a controlled cases )
* The Prospective Phase (600 patients who will be admitted and monitored in ICU in order to get at least 30 sepsis cases, according to our definition and criteria).

Measurements will be made from the forehead using the TTP's biocompatible sensor Unit that will be attached to the skin. The SU will transfer data to the MCU.

DETAILED DESCRIPTION:
TTP™ system, which is composed of 2 parts:

* SU - a disposable Sensor Unit patch
* MCU - e reusable Monitor Connecting Unit

The communication between the two units can be wired or wireless. The system to be used in this study is wired and the two units were connected via a Sensor Unit Cable (SCU).

The SU is attached to the temple area by a biocompatible disposable adhesive. It measures skin temperature across the temporal artery using several sensors, translates it to electrical signals and transmits those signals to the MCU. The MCU translates the electrical signals to core temperature using a special mathematical algorithm which overcomes the effect of the ambient temperature as well as the thermal properties of a specific patient. The core temperature as well as any concurrent error in the measurement process is displayed on the screen of the MCU or transmitted to the hospital VSM. The MCU has a wired connection to the hospital's VSM using Standard YSI400.

Study Objectives

The objectives of this clinical study are:

* A first objective of the clinical study is to verify the findings of a previously published study, relating to temperature pattern changes within patients who were diagnosed having sepsis , prior to its occurrence.
* A second objective is to examine the efficacy and safety of the TTP - a novel non-invasive core temperature measurement system , as a measure for continues core temperature monitoring.
* A third objective of the study, is to examine the effectiveness of the TTP as a measure for detection of temperature changes pattern and to correlate such changes with fever related to infections such as sepsis.

It is estimated that the study with take 18 months to complete.

Type of Study

* A Retrospective phase.
* A prospective phase

Temperature measurements Measurements will be made from the forehead using the TTP's biocompatible sensor Unit that will be attached to the skin The SU will transfer data to the MCU. The TTPTM system will be disinfected before use an alcohol-chlorhexidine solution.

1. The Retrospective Phase, screening temperature data logs of patients who had sepsis or other fever related infection. Screening period shall be at least 72 hours prior to sepsis or infection detection. This part shall include 50 sepsis cases and 30 non-sepsis cases as a control.
2. The Prospective Phase, measuring core temperature with the TTP and comparing it with existing technology such as rectal, esophageal or catheter or skin (by the case). The temperature data taken from each patient who will have a sepsis or other fever related infection will be analyzed to find any relation between the temperature pattern change Any medical care decision (such as microbiology cultures, additional testing, etc) will be made entirely according to existing reference standard of care. The TTP device will not influence in any way on ICU physician' decision. The TTP device purpose is only to record medical data for later evaluation and not to intertwine in medical care given to participants.

This part shall include up to 600 patients who will be monitored and analyzed during their stay in the ICU in order to get at least 30 sepsis cases.

ELIGIBILITY:
Study Participants - Patients hospitalized in ICU department.

Inclusion Criteria:

The Retrospective Phase

* Both genders (Male or Female).
* Aged 18 years and/or above.
* Patients were Admitted to our ICU for more than 3 days, and shall be at least 72 hours prior to sepsis or infection detection in the ICU The Prospective Phase

  * Both genders (Male or Female).
  * Aged 18 years and/or above. Patients expected to be admitted to our ICU for more than 3 days

Exclusion Criteria:

The patients will be excluded from the trial if one of the following occurs:

The Retrospective Phase

* No exclusion criteria The Prospective Phase

  - The medical staff decides that the patien t should not participate.
* Unavailable measurement site in case of head injury in the head area.
* Unavailable measurement reading during admission to ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Continuously measure body temperature using TTP | Estimated time frame of the trial is 18 months.
  During the trial, temperature measurements will be conducted using the TTP™ and currently used thermometers which are in routine use, later to be regarded as reference methods To examine the effectiveness of the TTP™ as a measure for detection of temperature changes pattern and to correlate such changes with fever related to infections such as sepsis.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No